CLINICAL TRIAL: NCT07298824
Title: Clinical Efficacy and Mechanism Exploration of MR-61 in Delaying the Progression of Myopia: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Clinical Efficacy and Mechanism Exploration of MR-61 in Delaying the Progression of Myopia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Yifeng Yu, Associate Chief Physician, Ph.D., Second Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IIT-I-2025-082
Record Dates: First submitted 2025-11-23; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Myopia Progressing
Keywords: Myopia,Probiotics,Gut microbiota
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): Oral administration of the investigational probiotic powder MR-61. The primary component is Bifidobacterium. Dosage: one sachet, 2-3 times daily, for 3 months.
  Interventions: Biological: Investigational Bifidobacterium Preparation MR-61
- Placebo group (Placebo Comparator): Oral administration of a matched placebo powder. Dosage: one sachet, 2-3 times daily, for 3 months.
  Interventions: Other: Placebo for MR-61

INTERVENTIONS:
Biological: Investigational Bifidobacterium Preparation MR-61 — Oral administration of the investigational probiotic powder MR-61. The primary component is Bifidobacterium. Dosage: one sachet, 2-3 times daily, for 3 months.
  Arms: Probiotic group
Other: Placebo for MR-61 — Oral administration of a matched placebo powder. Dosage: one sachet, 2-3 times daily, for 3 months.
  Arms: Placebo group

SUMMARY:
To investigate whether probiotic MR-61 can assist in slowing down the progression rate of myopia (a prospective randomized controlled study).

DETAILED DESCRIPTION:
To investigate whether probiotic MR-61 can assist in slowing down the progression rate of myopia (a prospective randomized controlled study).

ELIGIBILITY:
Inclusion Criteria:

1. Myopia is defined as spherical equivalent (SE) ≤ -0.5D.
2. Aged between 3 and 18 years, with no restriction on gender.
3. Cylinder power ≤ 1.50D; anisometropia of SE between both eyes ≤ 1.50D.
4. The subject has sufficient compliance with the study follow-up; the subject or their guardian has the intention to receive treatment and has signed the informed consent form.

Exclusion Criteria:

1. Presence of other concomitant ocular diseases;
2. Abnormal findings on clinical slit-lamp examination;
3. Existence of amblyopia, manifest strabismus, esotropia, or other congenital ocular diseases;
4. Individuals with abnormal intraocular pressure or abnormal axial length of the eye;
5. Either or both parents having a spherical equivalent (SE) ≤ -6.00D;
6. Other conditions inconsistent with this study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Spherical Equivalent Refraction | Measured at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  The change in spherical equivalent refraction (SER) from baseline to each follow-up visit, measured in diopters (D). SER is calculated as the spherical power plus half of the cylindrical power. A negative change indicates an increase in myopia.

SECONDARY OUTCOMES:
Change in Axial Length | Measured at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  The growth value of ocular axial length, measured in millimeters (mm).
Change in Corneal Curvature | Measured at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  The change in corneal curvature (keratometry), measured in diopters (D).
Change in Binocular Anisometropia | Measured at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  The difference in spherical equivalent refraction between the two eyes, measured in diopters (D).
Change in Anterior Chamber Depth | Measured at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  The change in depth of the anterior chamber of the eye, measured in millimeters (mm).
Change in Lens Thickness | Measured at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  The change in thickness of the crystalline lens, measured in millimeters (mm).
Change in Vitreous Cavity Depth | Measured at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  The change in depth of the vitreous cavity, measured in millimeters (mm)
Change in Far Phoria Degree | Measured at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  The degree of heterophoria for distance vision, measured in prism diopters (PD).
Change in Near Phoria Degree | Measured at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  The degree of heterophoria for near vision, measured in prism diopters (PD).
Score on the National Eye Institute Visual Function Questionnaire - 25 (NEI VFQ-25) | Assessed at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  Visual quality and vision-related quality of life is assessed using the National Eye Institute Visual Function Questionnaire - 25 (NEI VFQ-25). The overall composite score ranges from 0 to 100, where a higher score represents better visual function and quality of life.
Score on the Montreal Cognitive Assessment (MoCA) | Assessed at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  Cognitive function is assessed using the Montreal Cognitive Assessment (MoCA), a widely used screening test for cognitive impairment. The total score ranges from 0 to 30, with a score of 26 or higher considered normal. As probiotic supplementation may influence cognitive function, this will be considered in the interpretation of results.
Score on the Gastrointestinal Symptom Rating Scale (GSRS) | Assessed at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  Gastrointestinal symptoms are assessed using the Gastrointestinal Symptom Rating Scale (GSRS), a validated questionnaire covering reflux, abdominal pain, indigestion, diarrhea, and constipation. Each symptom is rated on a scale from 0 (no discomfort) to 6 (very severe discomfort). A higher total or subscale score indicates more severe gastrointestinal symptoms (worse outcome). As probiotic supplementation may influence gastrointestinal function, this will be considered in the interpretation of results.
Score on the World Health Organization Quality of Life Brief Version (WHOQOL-BREF) | Assessed at baseline, 1, 3, 6, 9, 12, 13, 14, 19, and 25 months post-intervention.
  Participant adaptation and overall quality of life are assessed using the World Health Organization Quality of Life Brief Version (WHOQOL-BREF), a validated generic quality of life instrument. It covers physical health, psychological health, social relationships, and environment domains. The total score is transformed to range from 0 to 100, where a higher score indicates a better quality of life and better adaptation. As probiotic supplementation may influence overall well-being, this will be considered in the interpretation of results.
Change in gut microbiota composition and diversity assessed by 16S rRNA gene sequencing | Fecal samples collected at baseline, 3, 6, 12, and 25 months post-intervention for sequencing analysis.
  Fecal samples collected before and after intervention are analyzed using full-length 16S rRNA gene sequencing. Key metrics include changes in alpha diversity indices (e.g., Shannon Index, observed species), beta diversity (e.g., weighted/unweighted UniFrac distance), and relative abundance of specific bacterial taxa (e.g., phylum Firmicutes/Bacteroidota ratio, genus Bifidobacterium).
Change in concentrations of fecal and serum metabolites | Fecal and blood serum samples collected at baseline, 3, 6, 12, and 25 months post-intervention for metabolite analysis.
  Targeted metabolomic analysis is performed on fecal and blood serum samples. Concentrations of specific metabolites (e.g., short-chain fatty acids, bile acids, or inflammatory cytokines) are measured and reported in nanomolar (nM) or picograms per milliliter (pg/mL) concentrations, as applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- Yifeng Yu, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided